CLINICAL TRIAL: NCT01527864
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Study to Evaluate the Efficacy of Paclitaxel-Carboplatin Alone or With Pegylated Endostatin for Advanced Non-small Cell Lung Cancer
Brief Title: Paclitaxel-Carboplatin Alone or With M2ES for Non-Small-Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Protgen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M2ES2011-1
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — CP protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pegylated endostatin (Experimental)
  Interventions: Drug: pegylated endostatin and Paclitaxel-Carboplatin
- Control (Placebo Comparator)
  Interventions: Drug: Placebo and Paclitaxel-Carboplatin

INTERVENTIONS:
Drug: pegylated endostatin and Paclitaxel-Carboplatin — Dosage：10mg/m2
  Other Names: M2ES
  Arms: pegylated endostatin
Drug: Placebo and Paclitaxel-Carboplatin — Dosage：10mg/m2
  Other Names: placebo
  Arms: Control

SUMMARY:
A phase II, multicenter, randomized, double-blind, placebo-controlled study was carried out. Patients were randomly assigned to the treatment (PC + pegylated endostatin) or the control group (PC+ placebo). The efficacy was evaluated every six weeks.Follow-up continued until disease progression or death.

DETAILED DESCRIPTION:
A randomized phase 2 study, involving patients with advanced non-small-cell lung cancer who had not previously received chemotherapy, compared paclitaxel and carboplatin Plus placebo with paclitaxel and carboplatin plus PEGylated endostatin, with PEGylated endostatin at a dose of 10 mg/m2 intravenously every weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, newly diagnosed stage IIIB or stage IV cancer or recurrent non-small-cell lung cancer for which they had not received chemotherapy, targeted therapy.
2. Prior radiation therapy was allowed provided that the only sites disease were not located in lung.
3. Measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST).
4. ≥18 years of age.
5. ECOG performance status of 0 or 1.
6. Life expectancy of at least 12 weeks.
7. Adequate hematologic, hepatic, and renal function.
8. Patients are voluntary to participate and sigh the informed contents.

Exclusion Criteria:

1. Major surgery within the prior 4 weeks.
2. Participating any clinical trial within the prior 4 weeks.
3. Patients had clinically apparent CNS disease ( primary brain tumors, tumor related apoplexy, CNS metastases, carcinomatous meningitis.)
4. Another active malignancy, or any history of other malignancy within the past 3 years except for nonmelanoma skin cancer and carcinoma in situ of the cervix.
5. Pregnant or lactating women.
6. Radiation therapy have not been completed 4 weeks before enrollment.
7. Pulmonary embolus, deep venous thrombosis or bleeding diathesis.
8. Uncontrolled intercurrent illness as following: prior or ongoing uncontrolled hypertension;angina pectoris; congestive cardiac failure; myocardial ischemia, infarction, uncompensated coronary artery disease within the past 12 months; Uncontrolled arrhythmia; Uncontrolled diabetes mellitus; Uncontrolled infection.
9. Grade 2 hemoptysis within the past 6 months.
10. Acute or chronic renal disease.
11. Active hepatitis or HIV.
12. ECG: QTC ≥ 480 ms.
13. Patients on therapeutic doses of heparin.
14. Other conditions that are regarded for exclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yan Sun, MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Cancer hospital, Chinese academy of medical science, Beijing, Beijing Municipality, China